CLINICAL TRIAL: NCT05777070
Title: Remote Ischemic Conditioning Combined With Bimanual Task Training to Enhance Bimanual Skill Learning and Corticospinal Excitability in Children With Unilateral Cerebral Palsy
Brief Title: Effects of Remote Ischemic Conditioning on Bimanual Skill Learning and Corticospinal Excitability in Children With Unilateral Cerebral Palsy
Acronym: RIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Carolina University (Other)
Responsible Party: Principal Investigator, Swati Manoharrao Surkar, Assistant Professor, East Carolina University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MS4_UMCIRB 21-001913
Record Dates: First submitted 2023-03-06; First posted 2023-03-20 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Unilateral Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Triple blinded, randomized controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants are masked to group assignments, investigators are masked to assessments, and outcomes assessors are masked to intervention groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote Ischemic Conditioning (RIC) (Experimental): RIC is achieved via blood pressure cuff inflation to at least 20 mmHg above systolic blood pressure to 250 mmHg on the more involved arm. RIC involves 5 cycles of 5 minutes blood pressure cuff inflation followed by alternating 5 minutes of cuff deflation and requires 45 minutes. RIC is performed on visits 1-7.
  Interventions: Behavioral: Bimanual Cup Stacking Training
- Sham conditioning (Sham Comparator): Sham conditioning is achieved via blood pressure cuff inflation to 25 mmHg on the more involved arm. RIC involves 5 cycles of 5 minutes blood pressure cuff inflation followed by alternating 5 minutes of cuff deflation and requires 45 minutes. RIC is performed on visits 1-7.
  Interventions: Behavioral: Bimanual Cup Stacking Training

INTERVENTIONS:
Behavioral: Bimanual Cup Stacking Training — Children practices bimanual cup stacking, 15 trials/day for 5 consecutive days
  Other Names: Remote limb ischemic conditioning; Sham conditioning

SUMMARY:
Unilateral cerebral palsy (UCP) is a leading cause of childhood disability. An early brain injury impairs the upper extremity function, bimanual coordination, and impacts the child's independence. The existing therapeutic interventions have higher training doses and modest effect sizes. Thus, there is a critical need to find an effective priming agent to enhance bimanual skill learning in children with UCP. This study aims to determine the effects of a novel priming agent, remote ischemic conditioning (RIC), when paired with bimanual skill training to enhance bimanual skill learning and to augment skill dependent plasticity in children with UCP.

DETAILED DESCRIPTION:
Ischemic conditioning (IC) is a phenomenon of protecting the target organ from ischemia by directly exposing it to brief episodes of sublethal ischemia. RIC is a clinically feasible way of performing IC where episodes of ischemia and reperfusion are delivered with cyclic inflation and deflation of a blood pressure cuff on the arm or leg. Pre-clinical and preliminary clinical trials in humans show neuroprotective effects of RIC. Investigators prior work has shown that when paired with motor training, RIC enhances motor learning in healthy individuals. Based on these diversified benefits of RIC, the central hypothesis is that the multifactorial mechanisms of RIC can be harnessed as a priming agent to enhance motor learning and augment neuroplasticity in children with UCP. The Specific Aims are: 1) to determine the effects of RIC + training on bimanual skill learning and bimanual coordination, and 2) to determine the effects of RIC + training on corticospinal excitability in children with UCP. In this triple blind, randomized controlled trial, 46 children with UCP, ages 6-16 years will first undergo bimanual speed stack performance, functional upper extremity, and Transcranial Magnetic Stimulation assessments. Children will then undergo RIC/Sham conditioning plus training. Investigators will deliver RIC/sham conditioning via cyclic inflation and deflation of a pressure cuff on the paretic arm using a standard protocol. Training will involve 5 days (15 trials/day) of bimanual speed stack training for 5 days. The children will perform the same baseline assessments post-intervention. Investigators hypothesize that compared to sham conditioning + training, RIC + training will significantly enhance: 1) bimanual skill performance (decrease in movement time (sec) to complete bimanual speed stack task), 2) bimanual coordination and bimanual function (improvement in kinematic variables and increase in the Assisting Hand Assessment scores), 3) cortical excitability in the ipsilesional primary motor cortex (M1) (larger amplitude of motor evoked potentials and lower resting or active motor thresholds), and 4) reduce motor cortex inhibition (reduced short-interval intracortical inhibition and increase in intracortical facilitation in ipsilesional M1). The long-term goal is to develop effective interventions to improve function of children with UCP. Outcomes of this project will provide critical ingredients for designing Phase II trials that will determine the effects of RIC combined with different dose of intensive behavioral interventions to improve functional outcomes in children with UCP.

ELIGIBILITY:
Inclusion Criteria:

1. Children diagnosed with unilateral cerebral palsy (UCP)
2. Manual Ability Classification System (MACS) levels I-III
3. Ability to complete a stack of 3 cups in 1 minute
4. Mainstream in school

Exclusion Criteria:

1. Children with other developmental disabilities such as autism, attention deficit hyperactivity disorder, developmental coordination disorders, etc.
2. Children with absent active motor threshold
3. Children with known cardiorespiratory, vascular, and metabolic disorders
4. Children with neoplasm and hydrocephalus
5. Children who are currently receiving or received other adjunct therapies such as rTMS and tDCS in the past 6 months
6. Children with seizures within last 2 years and on anti-seizure medications
7. Children with metal implants and incompatible medical devices

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Change in Bimanual Learning | Baseline and 1 week
  The time (seconds) to complete each trial of cup stack, which will be averaged across nine trials. This will be measured at visit 1 (pre-) and visit 7 (post-intervention).
Change in Symmetric performance and tangential velocities | Baseline and 1 week
  Symmetric performance is characterized as a time-lag between the affected and less affected arm during movement onset and task completion.
Change in Resting Motor Threshold (rMT) | Baseline and 1 week
  The rMT is the stimulator output required to produce a motor evoked potential (MEP) of > 50 μV in at least 5/10 trials in FDI muscle.
Change in Active Motor Threshold (aMT) | Baseline and 1 week
  The aMT is the stimulator output required to produce a motor evoked potential (MEP) of > 200 μV in FDI muscle during 30% of MVIC of FDI muscle using a pinch grip. aMT is a measure of motor cortex excitability.

SECONDARY OUTCOMES:
Change in Assisting Hand Assessment | Baseline and 1 week
  Assisting Hand Assessment assesses bimanual coordination and affected hand function. A 5-point change from pre- to post-intervention is considered a clinically meaningful improvement.
Change in Hand Trajectory | Baseline and 1 week
  Hand trajectory is defined as the resultant 3D path length between the starting position and task completion.
Change in Temporal coupling (normalized movement overlap time) | Baseline and 1 week
  Normalized movement overlap time is calculated as the percentage of total task completion time that both hands are participating in the stacking sequence during bimanual coordination task
Change in total participation time of each hand | Baseline and 1 week
  Total participation time is calculated as the total amount of time the affected and the less affected hand participate in bimanual coordination task. A hand will be considered as participating in the task any time the wrist marker tangential velocity remains over 2.0 cm/s for at least 100 ms.
Change in Goal Synchronization | Baseline and 1 week
  Goal synchronization is defined as a time lag between the initiation of the affected compared to the unaffected arm
Change in total task duration | Baseline and 1 week
  Total task duration is defined as the duration from movement onset until the criteria for task completion is reached with both hands.
Change in Stimulus response curve | Baseline and 1 week
  stimulus-response curves will be constructed for the ipsilesional as well as contralesional M1 at intensities of 90%, 100%, 110%, 120%, 130%, 140%, and 150% of rMT (10 stimuli per intensity in random order). The peak-to-peak amplitude of MEPs and area under the curve of resultant MEPs to these intensities will be calculated.
Change in Motor Evoked Potential (MEP) amplitude | Baseline and 1 week
  The peak-to-peak amplitude of the EMG response from the affected as well as unaffected FDI muscle while stimulating the ipsilesional as well as contralesional motor cortex will be recorded at 100% rMT and averaged across 10 single-pulse trials. MEP amplitude indicates the strength of motor response to TMS.
Change in Short-interval intracortical inhibition (SICI) and intracortical facilitation (ICF) | Baseline and 1 week
  SICI and ICF will be obtained by applying a conditioning stimulus at 80% rMT intensity or AMT intensity followed by a test stimulus at 120% rMT intensity over the hot spot. The interstimulus interval between the conditioning and test stimulus will be 3 ms for obtaining measures of SICI and 15 ms for obtaining ICF.

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Physical Therapy, East Carolina University, Greenville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared on NIH figshare network and will be made available on request.

REFERENCES:
- [Background] Kharbanda RK, Nielsen TT, Redington AN. Translation of remote ischaemic preconditioning into clinical practice. Lancet. 2009 Oct 31;374(9700):1557-65. doi: 10.1016/S0140-6736(09)61421-5. PMID 19880021
- [Result] Dirnagl U, Becker K, Meisel A. Preconditioning and tolerance against cerebral ischaemia: from experimental strategies to clinical use. Lancet Neurol. 2009 Apr;8(4):398-412. doi: 10.1016/S1474-4422(09)70054-7. PMID 19296922
- [Result] Gidday JM. Cerebral preconditioning and ischaemic tolerance. Nat Rev Neurosci. 2006 Jun;7(6):437-48. doi: 10.1038/nrn1927. PMID 16715053
- [Result] Stetler RA, Leak RK, Gan Y, Li P, Zhang F, Hu X, Jing Z, Chen J, Zigmond MJ, Gao Y. Preconditioning provides neuroprotection in models of CNS disease: paradigms and clinical significance. Prog Neurobiol. 2014 Mar;114:58-83. doi: 10.1016/j.pneurobio.2013.11.005. Epub 2014 Jan 2. PMID 24389580
- [Result] Mattlage AE, Sutter EN, Bland MD, Surkar SM, Gidday JM, Lee JM, Hershey T, Chen L, Lang CE. Dose of remote limb ischemic conditioning for enhancing learning in healthy young adults. Exp Brain Res. 2019 Jun;237(6):1493-1502. doi: 10.1007/s00221-019-05519-w. Epub 2019 Mar 26. PMID 30915491
- [Result] Sutter EN, Mattlage AE, Bland MD, Cherry-Allen KM, Harrison E, Surkar SM, Gidday JM, Chen L, Hershey T, Lee JM, Lang CE. Remote Limb Ischemic Conditioning and Motor Learning: Evaluation of Factors Influencing Response in Older Adults. Transl Stroke Res. 2019 Aug;10(4):362-371. doi: 10.1007/s12975-018-0653-8. Epub 2018 Aug 7. PMID 30088217
- [Result] Surkar SM, Bland MD, Mattlage AE, Chen L, Gidday JM, Lee JM, Hershey T, Lang CE. Effects of remote limb ischemic conditioning on muscle strength in healthy young adults: A randomized controlled trial. PLoS One. 2020 Feb 4;15(2):e0227263. doi: 10.1371/journal.pone.0227263. eCollection 2020. PMID 32017777
- [Derived] Surkar SM, Willson JD, Cassidy JM, Kantak S, Patterson CG. Remote ischaemic conditioning combined with bimanual task training to enhance bimanual skill learning and corticospinal excitability in children with unilateral cerebral palsy: a study protocol of a single centre, phase II randomised controlled trial. BMJ Open. 2023 Sep 28;13(9):e076881. doi: 10.1136/bmjopen-2023-076881. PMID 37770277